CLINICAL TRIAL: NCT03314688
Title: Lifestyle, Exercise, and Nutrition Study Early After Diagnosis (LEANer)
Brief Title: Lifestyle, Exercise, and Nutrition Study Early After Diagnosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2000020335; 1R01CA207753-01A1 (NIH)
Record Dates: First submitted 2017-09-13; First posted 2017-10-19 (Actual); Results first posted 2024-05-14 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Diet

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The following study personnel will be masked to participant study arm: the staff performing DXA scan and blood processing/biomarker evaluation. The staff performing clinic measures, study staff reviewing forms and entering data, the PI and Co-Is, the statistician, study manager, and interventionists (study dieticians) will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Group (Active Comparator): Standardized breast cancer follow up care and materials regarding treatment (i.e., chemotherapy and endocrine therapy when relevant).
  Lifestyle intervention books for breast cancer survivors at the end of the study. Women will also be offered a counselling session with a registered study dietician at the end of the study.
  Interventions: Behavioral: Usual Care
- Dietary/Physical Activity Intervention (Experimental): Eleven 30-min counseling sessions over six months (weekly, then biweekly, then monthly) with additional sessions in the latter 6 months (5 additional monthly sessions for a total of 16 sessions), timed with their oncology visit or via telephone if not coming in for oncology visit. Sessions focus on motivating health dietary choices and physical activity (home-based program).
  Interventions: Behavioral: Dietary/Physical Activity intervention

INTERVENTIONS:
Behavioral: Dietary/Physical Activity intervention — Motivational counseling to follow established dietary and exercise guidelines.
  Arms: Dietary/Physical Activity Intervention
Behavioral: Usual Care — Standard follow-up care and educational materials. Lifestyle counseling offered at the conclusion of the trial.
  Arms: Usual Care Group

SUMMARY:
The proposed study is a randomized trial evaluating the impact of a dietary and physical activity guidelines intervention vs. usual care on adherence to breast cancer treatments, body composition, and changes in biomarkers in 172 women newly diagnosed with breast cancer scheduled to receive neoadjuvant or adjuvant chemotherapy.

DETAILED DESCRIPTION:
Currently the Department of Health and Human Services, the American Cancer Society and others provide diet and exercise guidelines for cancer survivors. Many women with breast cancer do not follow these guidelines, and also elect to delay concerted efforts toward following them until active treatment is complete. However, adoption of these recommended lifestyle behaviors soon after diagnosis may prevent adverse changes in body composition and breast cancer biomarkers and may even improve the efficacy of treatment resulting in improved breast cancer prognosis. Further, by increasing our understanding of the mechanisms mediating the association between lifestyle behaviors and breast cancer survival, this study will improve our knowledge of how changes in diet and physical activity influence breast cancer outcomes. Lastly, guidelines for breast cancer survivors also overlap with those for diabetes and cardiovascular disease (CVD) prevention, the latter being a common cause of breast cancer mortality.

The proposed study will examine, in 172 women newly diagnosed with Stage I-III breast cancer who are not practicing the dietary and lifestyle guidelines, and who are scheduled to receive neoadjuvant or adjuvant chemotherapy, the effect of a 1-year dietary and physical activity guidelines intervention vs. usual care on the following breast cancer outcomes measured before beginning chemotherapy (Time 0), post chemotherapy (Time 1), at one-year post-diagnosis (Time 2), at two years post-diagnosis (Time 3), and at five-years post-diagnosis (Time 4): adherence to treatment, and changes in biomarkers, body composition, diet, physical activity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Stage I-III breast cancer
* Scheduled to receive neoadjuvant or adjuvant chemotherapy
* Physically able to walk
* Able to complete forms, understand instructions and read intervention book in English
* Agrees to be randomly assigned to either intervention or usual care group

Exclusion Criteria:

* Women who have completed their 2nd chemotherapy
* Women already practicing dietary or physical activity guidelines
* Are pregnant or intending to become pregnant in the next year
* Recent (past year) stroke/myocardial infarction or congestive heart failure/ejection fraction < 40%
* Presence of dementia or major psychiatric disease
* Non-English speaking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2026-07-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Irwin, Ph.D., Principal Investigator — Yale University; Tara Sanft, M.D., Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - Dana Farber Cancer Center, Boston, Massachusetts

REFERENCES:
- [Derived] Puklin LS, Li FY, Ferrucci LM, Cartmel B, Harrigan M, McGowan C, Zupa M, Ligibel JA, Sanft T, Irwin ML. Effect of a lifestyle intervention during chemotherapy for breast cancer on quality of life. JNCI Cancer Spectr. 2026 Jan 9;10(1):pkaf125. doi: 10.1093/jncics/pkaf125. PMID 41452765
- [Derived] Sanft T, Harrigan M, McGowan C, Cartmel B, Zupa M, Li FY, Ferrucci LM, Puklin L, Cao A, Nguyen TH, Neuhouser ML, Hershman DL, Basen-Engquist K, Jones BA, Knobf T, Chagpar AB, Silber A, Tanasijevic A, Ligibel JA, Irwin ML. Randomized Trial of Exercise and Nutrition on Chemotherapy Completion and Pathologic Complete Response in Women With Breast Cancer: The Lifestyle, Exercise, and Nutrition Early After Diagnosis Study. J Clin Oncol. 2023 Dec 1;41(34):5285-5295. doi: 10.1200/JCO.23.00871. Epub 2023 Sep 1. PMID 37656930
- [Derived] Sanft T, Harrigan M, Cartmel B, Ferrucci LM, Li FY, McGowan C, Zupa M, Nguyen TH, Ligibel J, Neuhouser ML, Hershman DL, Basen-Engquist K, Jones B, Knobf T, Chagpar A, Silber A, Irwin ML. Effect of healthy diet and exercise on chemotherapy completion rate in women with breast cancer: The Lifestyle, Exercise and Nutrition Early after Diagnosis (LEANer) study: Study protocol for a randomized clinical trial. Contemp Clin Trials. 2021 Oct;109:106508. doi: 10.1016/j.cct.2021.106508. Epub 2021 Jul 16. PMID 34274495

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care Group: Standardized breast cancer follow up care and materials regarding treatment (i.e., chemotherapy and endocrine therapy when relevant).
  Lifestyle intervention books for breast cancer survivors at the end of the study. Women will also be offered a counselling session with a registered study dietician at the end of the study.
  Usual Care: Standard follow-up care and educational materials. Lifestyle counseling offered at the conclusion of the trial.
Period: Overall Study
Arm/Group | Dietary/Physical Activity Intervention | Usual Care Group
Started | 87 | 86
Eligible for Endocrine Therapy | 40 | 37
Completed | 87 | 86
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dietary/Physical Activity Intervention | Usual Care Group | Total
Number analyzed (Participants) | 87 | 86 | 173
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (11.3) | 53.3 (10.9) | 52.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 86 | 173
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race and Ethnicity: Non-Hispanic White | 61 | 62 | 123
  Race and Ethnicity: Non-Hispanic Black | 11 | 14 | 25
  Race and Ethnicity: Hispanic | 8 | 5 | 13
  Race and Ethnicity: Asian or Pacific Islander | 2 | 4 | 6
  Race and Ethnicity: Prefer not to answer | 3 | 0 | 3
  Race and Ethnicity: Other | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 87 | 86 | 173
Study Site [Count of Participants; unit: Participants]
  Yale | 63 | 59 | 122
  Dana-Farber Cancer Institute | 24 | 27 | 51
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.5 (7.0) | 29.8 (6.6) | 29.7 (6.8)
Postmenopausal Status [Count of Participants; unit: Participants]
  Postmenopausal: Yes | 48 | 46 | 94
  Postmenopausal: No | 39 | 40 | 79
Cancer Stage [Count of Participants; unit: Participants] — This measure is from the five stages of breast cancer, starting at zero and going up to four. Stages are represented by the Roman numerals I, II, III, and IV. Stage IV is the most advanced stage of breast cancer.
  Participants
    Stage I | 45 | 43 | 88
    Stage II | 31 | 34 | 65
    Stage III | 11 | 9 | 20
Receptor Status [Count of Participants; unit: Participants]
  ER/PR+, HER2- | 49 | 50 | 99
  ER/PR+/-, HER2+ | 15 | 15 | 30
  Triple negative | 23 | 21 | 44
Chemotherapy [Count of Participants; unit: Participants]
  Neoadjuvant | 41 | 32 | 73
  Adjuvant | 46 | 54 | 100
Chemotherapy Cycles [Count of Participants; unit: Participants]
  4 (range of weeks: 8-12) | 23 | 25 | 48
  >4 (range of weeks: 12-24) | 64 | 61 | 125
Time since diagnosis [Mean (Standard Deviation); unit: days] | 60 (34) | 68 (32) | 63 (33)

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Treatment Measured by Chemotherapy Completion Rate
Description: Chemotherapy completion rate will be assessed (via medical records) as the average relative dose-intensity (RDI) for the originally planned regimen based on standard formulas. RDI is calculated by dividing the participant's actual dose by the planned dose to get a percentage of actual dose/planned dose.
Time Frame: before initiating chemotherapy to post-chemotherapy, up to 7 months
Measure: Mean (Standard Deviation); unit: percentage of actual dose/planned dose
Arm/Group | Dietary/Physical Activity Intervention | Usual Care Group
Number analyzed (Participants) | 87 | 86
percentage of actual dose/planned dose | 93.9 (12.1) | 93.6 (11.1)
Statistical Analysis 1: Comparison: Dietary/Physical Activity Intervention vs Usual Care Group; Test type: Superiority; p = 0.69, t-test, 2 sided

2. Primary Outcome: Adherence to Endocrine Therapy in Women Taking Tamoxifen or Aromatase Inhibitors (AIs)
Description: This outcome was updated when results were entered. COVID restrictions prevented the intended method of assessment using urine collection. In its place are the responses on 3 questions regarding adherence.
  1. In the past month, how often did you take your aromatase inhibitor (AI)/tamoxifen pills as the doctor prescribed? ('All the time' responses counted)
  2. In the past month, how often did you forget to take one or more of your aromatase inhibitor (AI)/tamoxifen pills? ('Never' responses counted)
  3. In the past month, how often did you decide to skip one or more of your aromatase inhibitor (AI)/tamoxifen pills? ('Never' responses counted)
Time Frame: 12 months after enrollment
Population: Participants eligible for Endocrine Therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Dietary/Physical Activity Intervention | Usual Care Group
Number analyzed (Participants) | 40 | 37
Participants
  Q1. All the Time | 29 | 23
  Q2. Never | 23 | 18
  Q3. Never | 35 | 29
Statistical Analysis 1: Comparison: Dietary/Physical Activity Intervention vs Usual Care Group; Comparison of Q1: In the past month, how often did you take your aromatase inhibitor (AI)/tamoxifen pills as the doctor prescribed? = 'All the time'; Test type: Superiority; p = 0.33, Chi-squared
Statistical Analysis 2: Comparison: Dietary/Physical Activity Intervention vs Usual Care Group; Comparison of Q2: In the past month, how often did you forget to take one or more of your aromatase inhibitor (AI)/tamoxifen pills? = 'Never'; Test type: Superiority; p = 0.44, Chi-squared
Statistical Analysis 3: Comparison: Dietary/Physical Activity Intervention vs Usual Care Group; Comparison of Q3: In the past month, how often did you decide to skip one or more of your aromatase inhibitor (AI)/tamoxifen pills? = 'Never'; Test type: Superiority; p = 0.29, Chi-squared

3. Primary Outcome: Adherence to Endocrine Therapy in Women Taking Tamoxifen or Aromatase Inhibitors (AIs).
Description: This outcome was updated when results were entered. COVID restrictions prevented the intended method of assessment using urine collection. In its place are the responses on 3 questions regarding adherence.
  In the past month, how often did you take your aromatase inhibitor (AI)/tamoxifen pills as the doctor prescribed? ('All the time' responses counted- Q1) In the past month, how often did you forget to take one or more of your aromatase inhibitor (AI)/tamoxifen pills? ('Never' responses counted- Q2) In the past month, how often did you decide to skip one or more of your aromatase inhibitor (AI)/tamoxifen pills? ('Never' responses counted- Q3)
Time Frame: 24 months after enrollment
Population: Participants eligible for Endocrine Therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Dietary/Physical Activity Intervention | Usual Care Group
Number analyzed (Participants) | 40 | 37
Participants
  Q1. = All the Time | 22 | 22
  Q2. = Never | 20 | 18
  Q3. = Never | 33 | 25
Statistical Analysis 1: Comparison: Dietary/Physical Activity Intervention vs Usual Care Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.69, Chi-squared
Statistical Analysis 2: Comparison: Dietary/Physical Activity Intervention vs Usual Care Group; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.91, Chi-squared
Statistical Analysis 3: Comparison: Dietary/Physical Activity Intervention vs Usual Care Group; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.13, Chi-squared

4. Secondary Outcome: Pathological Complete Response
Description: In the subset of patients receiving neoadjuvant chemotherapy, no evidence of viable invasive tumor cells at the primary tumor site and axillary lymph nodes in the surgical specimen.
Time Frame: At the time of surgical resection following initial course of chemotherapy
Reporting Status: Not Posted

5. Secondary Outcome: Insulin Level
Description: Assessed by fasting blood (fast of 12 hours or more).
Time Frame: Baseline (pre-chemotherapy)
Reporting Status: Not Posted

6. Secondary Outcome: Insulin Level
Description: Assessed by fasting blood (fast of 12 hours or more).
Time Frame: Up to 7 months from treatment onset
Reporting Status: Not Posted

7. Secondary Outcome: Insulin Level
Description: Assessed by fasting blood (fast of 12 hours or more).
Time Frame: one year post-diagnosis
Reporting Status: Not Posted

8. Secondary Outcome: Insulin Level
Description: Assessed by fasting blood (fast of 12 hours or more).
Time Frame: two years post-diagnosis
Reporting Status: Not Posted

9. Secondary Outcome: C-reactive Protein Level
Description: Assessed by fasting blood (fast of 12 hours or more).
Time Frame: Baseline (pre-chemotherapy)
Reporting Status: Not Posted

10. Secondary Outcome: C-reactive Protein Level
Description: Assessed by fasting blood (fast of 12 hours or more).
Time Frame: Up to 7 months from treatment onset
Reporting Status: Not Posted

11. Secondary Outcome: C-reactive Protein Level
Description: Assessed by fasting blood (fast of 12 hours or more).
Time Frame: one year post-diagnosis
Reporting Status: Not Posted

12. Secondary Outcome: C-reactive Protein Level
Description: Assessed by fasting blood (fast of 12 hours or more).
Time Frame: two years post-diagnosis
Reporting Status: Not Posted

13. Secondary Outcome: Body Composition-body Weight
Description: Assessed by measured weight
Time Frame: Baseline (pre-chemotherapy)
Reporting Status: Not Posted

14. Secondary Outcome: Body Composition-body Mass Index (BMI)
Description: Assessed from measured weight and measured height
Time Frame: Baseline (pre-chemotherapy)
Reporting Status: Not Posted

15. Secondary Outcome: Body Composition-body Fat
Description: Assessed by dual energy X-ray absorptiometry (DEXA)
Time Frame: Baseline (pre-chemotherapy)
Reporting Status: Not Posted

16. Secondary Outcome: Body Composition-lean Body Mass
Description: Assessed by dual energy X-ray absorptiometry (DEXA)
Time Frame: Baseline (pre-chemotherapy)
Reporting Status: Not Posted

17. Secondary Outcome: Body Composition-bone Mineral Density
Description: Assessed by dual energy X-ray absorptiometry (DEXA)
Time Frame: Baseline (pre-chemotherapy)
Reporting Status: Not Posted

18. Secondary Outcome: Body Composition-body Weight
Description: Assessed by measured weight
Time Frame: Up to 7 months from treatment onset
Reporting Status: Not Posted

19. Secondary Outcome: Body Composition-body Mass Index (BMI)
Description: Assessed from measured weight and measured height
Time Frame: Up to 7 months from treatment onset
Reporting Status: Not Posted

20. Secondary Outcome: Body Composition-body Fat
Description: Assessed by dual energy X-ray absorptiometry (DEXA)
Time Frame: Up to 7 months from treatment onset
Reporting Status: Not Posted

21. Secondary Outcome: Body Composition-lean Body Mass
Description: Assessed by dual energy X-ray absorptiometry (DEXA)
Time Frame: Up to 7 months from treatment onset
Reporting Status: Not Posted

22. Secondary Outcome: Body Composition-bone Mineral Density
Description: Assessed by dual energy X-ray absorptiometry (DEXA)
Time Frame: Up to 7 months from treatment onset
Reporting Status: Not Posted

23. Secondary Outcome: Body Composition-body Weight
Description: Assessed by measured weight
Time Frame: one year post-diagnosis
Reporting Status: Not Posted

24. Secondary Outcome: Body Composition-BMI
Description: Assessed from measured weight and measured height
Time Frame: one year post-diagnosis
Reporting Status: Not Posted

25. Secondary Outcome: Body Composition-body Fat
Description: Assessed by dual energy X-ray absorptiometry (DEXA)
Time Frame: one year post-diagnosis
Reporting Status: Not Posted

26. Secondary Outcome: Body Composition-lean Body Mass
Description: Assessed by dual energy X-ray absorptiometry (DEXA)
Time Frame: one year post-diagnosis
Reporting Status: Not Posted

27. Secondary Outcome: Body Composition-bone Mineral Density.
Description: Assessed by dual energy X-ray absorptiometry (DEXA)
Time Frame: one year post-diagnosis
Reporting Status: Not Posted

28. Secondary Outcome: Body Composition-body Weight
Description: Assessed by measured weight
Time Frame: two years post-diagnosis
Reporting Status: Not Posted

29. Secondary Outcome: Body Composition-BMI
Description: Assessed from measured weight and measured height
Time Frame: two years post-diagnosis
Reporting Status: Not Posted

30. Secondary Outcome: Body Composition-body Fat
Description: Assessed by dual energy X-ray absorptiometry (DEXA)
Time Frame: two years post-diagnosis
Reporting Status: Not Posted

31. Secondary Outcome: Body Composition-lean Bone Mass
Description: Assessed by dual energy X-ray absorptiometry (DEXA)
Time Frame: two years post-diagnosis
Reporting Status: Not Posted

32. Secondary Outcome: Body Composition-bone Mineral Density
Description: Assessed by dual energy X-ray absorptiometry (DEXA)
Time Frame: two years post-diagnosis
Reporting Status: Not Posted

33. Secondary Outcome: Quality of Life
Description: Measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) questionnaire.
Time Frame: Baseline (pre-chemotherapy)
Reporting Status: Not Posted

34. Secondary Outcome: Quality of Life
Description: Measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) questionnaire.
Time Frame: Up to 7 months from treatment onset
Reporting Status: Not Posted

35. Secondary Outcome: Quality of Life
Description: Measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) questionnaire.
Time Frame: one year post-diagnosis
Reporting Status: Not Posted

36. Secondary Outcome: Quality of Life
Description: Measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) questionnaire.
Time Frame: two years post-diagnosis
Reporting Status: Not Posted

37. Secondary Outcome: Fecal Microbiome
Description: Assessed by stool collection.
Time Frame: Baseline (pre-chemotherapy)
Reporting Status: Not Posted

38. Secondary Outcome: Fecal Microbiome
Description: Assessed by stool collection.
Time Frame: Up to 7 months from treatment onset
Reporting Status: Not Posted

39. Secondary Outcome: Fecal Microbiome
Description: Assessed by stool collection.
Time Frame: one year post-diagnosis
Reporting Status: Not Posted

40. Secondary Outcome: Fecal Microbiome
Description: Assessed by stool collection.
Time Frame: two years post-diagnosis
Reporting Status: Not Posted

41. Secondary Outcome: Healthy Eating Index
Description: Assessed by food frequency questionnaire
Time Frame: five years post-diagnosis
Reporting Status: Not Posted

42. Secondary Outcome: Minutes Per Week of Moderate/Vigorous Physical Activity
Description: Assessed by the modified physical activity questionnaire
Time Frame: five years post-diagnosis
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 24 months
Description: PRO-CTCAE was used to assess participant Adverse Events.
Groups:
- Usual Care Group: Standardized breast cancer follow up care and materials regarding treatment (i.e., chemotherapy and endocrine therapy when relevant).
  Lifestyle intervention books for breast cancer survivors at the end of the 2-year study. Women will also be offered a counselling session with a registered study dietician at the end of the study.
  Usual Care: Standard follow-up care and educational materials. Lifestyle counseling offered at the conclusion of the trial.
Arm/Group | Dietary/Physical Activity Intervention | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 0/87 | 5/86
Serious Adverse Events (participants affected / at risk) | 45/87 | 47/86
Other Adverse Events (participants affected / at risk) | 78/87 | 70/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Dietary/Physical Activity Intervention (N=87) | Usual Care Group (N=86)
Severity of dry mouth (Gastrointestinal disorders) | 14/82 | 14/74
Severity of difficulty swallowing (Gastrointestinal disorders) | 2/82 | 6/74
Severity of mouth or throat sores (Infections and infestations) | 4/82 | 5/74
Inference of mouth or throat sores (Infections and infestations) | 1/82 | 5/74
Severity of problems with tasting (Nervous system disorders) | 17/82 | 16/74
Severity of decreased appetite (Metabolism and nutrition disorders) | 14/82 | 7/74
Inference of decreased appetite (Metabolism and nutrition disorders) | 7/82 | 7/74
Frequency of nausea (Gastrointestinal disorders) | 10/82 | 7/74
Severity of nausea (Gastrointestinal disorders) | 8/82 | 5/74
Severity of vomiting (Gastrointestinal disorders) | 1/82 | 2/74
Frequency of heartburn (Gastrointestinal disorders) | 13/82 | 13/74
Severity of heartburn (Gastrointestinal disorders) | 8/82 | 7/74
Severity of constipation (Gastrointestinal disorders) | 12/82 | 9/74
Frequency of diarrhea (Gastrointestinal disorders) | 13/82 | 12/74
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Dietary/Physical Activity Intervention (N=87) | Usual Care Group (N=86)
Severity of dry mouth (Gastrointestinal disorders) | 46/82 | 44/74
Severity of difficulty swallowing (Gastrointestinal disorders) | 23/82 | 20/74
Severity of mouth or throat sores (Infections and infestations) | 31/82 | 30/74
Inference of mouth or throat sores (Infections and infestations) | 15/82 | 19/74
Severity of problems with tasting (Nervous system disorders) | 58/82 | 52/74
Severity of decreased appetite (Metabolism and nutrition disorders) | 39/82 | 39/74
Inference of decreased appetite (Metabolism and nutrition disorders) | 24/82 | 27/74
Frequency of nausea (Gastrointestinal disorders) | 41/82 | 28/74
Severity of nausea (Gastrointestinal disorders) | 40/82 | 21/74
Frequency of vomiting (Gastrointestinal disorders) | 10/82 | 5/74
Severity of vomiting (Gastrointestinal disorders) | 8/82 | 6/74
Frequency of heartburn (Gastrointestinal disorders) | 41/82 | 37/74
Severity of heartburn (Gastrointestinal disorders) | 34/82 | 31/74
Severity of constipation (Gastrointestinal disorders) | 32/82 | 25/74
Frequency of diarrhea (Gastrointestinal disorders) | 41/82 | 33/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-14): https://cdn.clinicaltrials.gov/large-docs/88/NCT03314688/Prot_SAP_001.pdf
  • Informed Consent Form (2021-02-04): https://cdn.clinicaltrials.gov/large-docs/88/NCT03314688/ICF_000.pdf